CLINICAL TRIAL: NCT05999565
Title: Investigation of the Effect of Motor Imagery Training on Pain, Pain Beliefs, Functional Status and Neck Awareness in Individuals with Cervical Discogenic Pain
Brief Title: Investigation of the Effect of Motor Imagery Training in Individuals with Cervical Discogenic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, T Dere, Yozgat Bozok Unıversity, Hacettepe University
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tugbadere
Record Dates: First submitted 2023-07-22; First posted 2023-08-21 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-07

CONDITIONS: Image, Body; Neck Pain; Disc Herniation
Keywords: imagery; neck pain; disc herniation; exercise training; awareness
MeSH Terms: conditions — Neck Pain; Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Motor Imagery Training (Experimental): Motor Imagery Training Motor Imagery Training will be applied only to the 2nd group, under the supervision of a physiotherapist, twice a week for 8 weeks, for 20 minutes each session. The treatment duration for the 2nd group will be planned to be a total of 50 minutes, including both motor imagery and motor control exercises. Motor imagery sessions will take place in a quiet environment, with individuals comfortably seated.
  Lateralization Training Kinesthetic Imagery Visual Imagery Mirror-Image Active Exercise: Between weeks 6 and 8 of motor imagery training, the active exercises (Stretching Exercises, Active Exercises, and Endurance Exercises) will be actively performed in front of a mirror
  Interventions: Other: Motor Imagery Exercises; Other: Motor Control Exercises
- Motor Control Exercise (Experimental): Stretching Exercises: Stretching exercises will be applied to the cervical muscles, pectoral muscles, back, and shoulder muscles. Individuals will be asked to perform flexion, extension, lateral flexion, and rotational normal joint movements in the cervical region, and hold the end position for a few seconds. All stretching exercises will be performed for 15 repetitions.
  Active Exercises: To strengthen the cervical muscle groups, individuals will be taught how to use a mild to moderate resistance theraband for cervical flexion, extension, and lateral flexion, without compromising the chin tuck movement. Each movement will be performed for 10 repetitions, with 5-second rest intervals between exercises.
  Endurance Exercises: Before starting the endurance exercises, individuals will be taught the contraction of deep cervical flexors to gain automatic postural stabilization, and they will be instructed to maintain this movement in every exercise and activity.
  Interventions: Other: Motor Control Exercises

INTERVENTIONS:
Other: Motor Imagery Exercises — Lateralization Training: Individuals with cervical discogenic pain will receive lateralization training using a mobile application called "Recognize Neck" from the Neuro Orthopaedic Institute in Adelaide, Australia.
  Kinesthetic Imagery: During this training, individuals will be asked to actively perform exercises and feel the movements. In a quiet environment, a therapist will verbally describe the exercises, and individuals will be asked to imagine the positions of their bodies, the surface they are on, and the desired postures.
  Visual Imagery: Individuals will be asked to actively perform exercises and visualize the movements. In a quiet environment, a therapist will verbally describe the exercises, and individuals will be asked to mentally visualize their body positions, the surface they are on, and the exercises.
  Mirror-Image Active Exercise: Between weeks 6 and 8 of motor imagery training, the active exercises in front of a mirror.
  Arms: Motor Imagery Training
Other: Motor Control Exercises — Stretching Exercises: Stretching exercises will be applied to the cervical muscles, pectoral muscles, back, and shoulder muscles. Individuals will be asked to perform flexion, extension, lateral flexion, and rotational normal joint movements in the cervical region, and hold the end position for a few seconds. All stretching exercises will be performed for 15 repetitions.
  Active Exercises: To strengthen the cervical muscle groups, individuals will be taught how to use a mild to moderate resistance theraband for cervical flexion, extension, and lateral flexion, without compromising the chin tuck movement. Each movement will be performed for 10 repetitions, with 5-second rest intervals between exercises.
  Endurance Exercises: Before starting the endurance exercises, individuals will be taught the contraction of deep cervical flexors to gain automatic postural stabilization, and they will be instructed to maintain this movement in every exercise and activity.

SUMMARY:
In this study, motor control exercises including cervical region, upper extremity and scapular region muscles will be applied routinely in individuals with chronic neck pain. The application will been investigating, called motor imagery training, will been carried out together with motor control exercises.

DETAILED DESCRIPTION:
This training is a mental exercise method based on imagining exercises that are performed actively without any interventional application inside or outside the body, in a comfortable environment and without fatigue. It is thought that motor imagery training applied together with motor control exercises will contribute to the management of chronic neck pain due to cervical disc herniation and symptoms related to pain.

All individuals with cervical discogenic pain who met the inclusion criteria were assigned to '1. Group' and '2. It will be divided into two groups. It is planned to include approximately 20 individuals with cervical discogenic pain in each group. The sample size of the study will be determined by the power analysis to be made as a result of the pilot study to be carried out on 10 patients with the support of Biostatistics USA.

Group 1: (estimated) 20 Individuals with Cervical Discogenic Pain Group 2: (estimated) 20 Individuals with Cervical Discogenic Pain

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 65,
* Having a diagnosis of cervical disc herniation based on MRI findings, clinical, and physical examination,
* Experiencing neck pain for 3 months or longer,
* Having a resting pain intensity rated 3-7 (moderate severity) on the "Visual Analog Scale" for pain assessment (36),
* Classifying neck pain according to the 'Neck Pain Task Force' clinical classification system as Grade 3 (neck pain with accompanying neurological symptoms) or above,
* Having a Mini-Mental Test score of 24 or higher for the evaluation of cognitive functions.

Exclusion Criteria:

* Having a history of spinal tumor, spinal deformities, congenital malformation, or head trauma,
* Undergoing cervical spine surgery in the last 6 months,
* Having a presence of systemic, cardiorespiratory, central nervous system, or rheumatic diseases, any musculoskeletal or craniocervical disorders, or a history of headache.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of Normal Joint Range of Motion | September 2023-July 2024 (11 months)
  The cervical region and upper extremity normal range of motion of individuals with cervical discogenic pain will be evaluated using a universal goniometer.
Evaluation of Pain | september 2023-july 2024(11 months)
  In order to evaluate the pain levels of individuals with cervical disc herniation, the 10 cm Visual Analog Scale (VAS) developed by Price et al. to evaluate the level of pain in individuals with chronic pain will be used. 0; No pain, 10; means the most severe pain and individuals will be asked to indicate their neck pain level on the line.
Evaluation of Pain | september 2023-july 2024(11 months)
  Algometer Device (Baseline Push-Pull Force Gauge®, Fabrication Enterprises, Inc) will be used to evaluate the pain threshold in the individuals included in the study
Assessment of Pain-Related Beliefs | september 2023-july 2024(11 months)
  Pain Catastrophizing Scale Fear Avoidance Beliefs Questionnaire Pain Beliefs Questionnaire
Evaluation of Functional Status 1 | september 2023-july 2024(11 months)
  Assessment of Neck Disability; The Neck Disability Index
Evaluation of Functional Status 2 | september 2023-july 2024(11 months)
  Assessment of Muscle Strength: To evaluate the cervical and upper extremity muscle strength of individuals with cervical discogenic pain, measurements will be taken during maximum voluntary isometric contractions
Evaluation of Functional Status 3 | september 2023-july 2024(11 months)
  Assessment of Muscle Endurance: Neck Flexor Muscles, Neck Deep Flexor Muscles, Neck Extensor Muscles
Evaluation of Functional Status 4 | september 2023-july 2024(11 months)
  Assessment of Upper Extremity Functionality: The Nine-Hole Peg Test will be used to evaluate the upper extremity functionality of the individuals
Evaluation of Functional Status 5 | september 2023-july 2024(11 months)
  Upper Extremity Functional Index-15
Examination of Pathological Changes in the Disc | september 2023-july 2024(11 months)
  Examination of Pathological Changes in the Disc In our study, Magnetic Resonance Imaging (MRI) will be used to determine the structure of the disc and the severity of herniation. MRI is a non-invasive assessment method for examining disc herniation and identifying pathological changes in the disc. With MRI, various parameters will be examined, such as bulging, disc protrusion, disc extrusion, disc sequestration, central/paracentral, posterolateral disc herniation, nerve root compression, and disc degeneration. MRI evaluations will be performed using T2 and T1-weighted sagittal sections and T2-weighted axial sections as references. The anterior-posterior (AP) disc height and herniation thickness from the midpoint of the AP length will be evaluated in millimeters (mm).
Motor Imagery Ability Assessment 1 | september 2023-july 2024(11 months)
  The Motor Imagery Questionnaire-3 (MIQ-3) is used to assess motor imagery ability. It is designed to evaluate individuals' capacity to mentally simulate and visualize movements in their minds. MIQ-3 is commonly used among athletes, dancers, and individuals engaged in various physical activities.
Motor Imagery Ability Assessment 2 | september 2023-july 2024(11 months)
  Mental Chronometry is a method used to measure the time it takes for individuals to mentally process and execute specific movements or tasks in their minds. It provides insights into the speed and accuracy of mental movement representations.
Motor Imagery Ability Assessment 3 | september 2023-july 2024(11 months)
  Lateralization Test is employed to determine the degree of lateralization in individuals, specifically assessing their preference for using one side of the body over the other. It helps to understand the dominance of the left or right hemisphere of the brain in controlling motor functions.
Neck Awareness Assessment | september 2023-july 2024(11 months)
  The Fremantle Neck Awareness Questionnaire will be used to assess the level of neck awareness in the individuals included in the study.
  For the assessment of neck proprioception awareness, the cervical range of motion (CROM) device (Performance Attainment Associates, St. Paul, Minnesota, 55117, United States) will be used.
Evaluation of Movement Fear | september 2023-july 2024(11 months)
  The movement fears of the included participants will be assessed using the Tampa Scale for Kinesiophobia (TSK), developed by Kori et al.
Evaluation of Avoidance Behavior | september 2023-july 2024(11 months)
  For evaluating avoidance behavior due to pain, the Fear-Avoidance Component Scale will be used.
Evaluation of Participant Satisfaction | september 2023-july 2024(11 months)
  For assessing the satisfaction rate of individuals with cervical discogenic pain during the treatment period, the Short Form of Patient Satisfaction Assessment will be used. The form was developed by Hawthorne et al. in 2006, and its Turkish validity has been established by Şen et al. The scale consists of the following scoring criteria: for items 1, 2, 4, and 7: 0=Very satisfied, 1=Satisfied, 2=Neither satisfied nor dissatisfied, 3=Dissatisfied, 4=Very dissatisfied; for items 3 and 6: 0=Strongly agree, 1=Agree, 2=Undecided, 3=Disagree, 4=Strongly disagree, and item 5 is scored as 0=Always, 1=Most of the time, 2=Half of the time, 3=Sometimes, 4=Never. For scoring item 6, it needs to be reversed. The total score obtained from the scale is interpreted as follows: 0-10 points indicate very satisfied, 11-18 points indicate satisfied, 19-26 points indicate dissatisfied, and 27-28 points indicate very dissatisfied. An increase in scores signifies an increase in dissatisfaction level
Evaluation of Participants' Views on the Treatment | september 2023-july 2024(11 months)
  The views of individuals with cervical discogenic pain regarding the treatment will be assessed through a specially prepared form for this study. The form includes a total of 5 open-ended questions, addressing the participants' opinions on the treatment they received. Participants will be asked to verbally respond to questions about the changes they observed after the treatment, the contributions of the treatment, the easiest or most challenging aspects of the treatment, and whether they would like to continue with this treatment. The responses of participants to the open-ended questions will be recorded using an audio recording system, and later, the evaluator will listen to the recording and transcribe all the answers in written form.

CONTACTS AND LOCATIONS:
Overall Officials: İpek GÜRBÜZ, PT, Prof, Study Director — Hacettepe University
Locations (2):
- Turkey (Türkiye) (2):
  - School of Sarıkaya Physical Therapy and Rehabilitation, Yozgat
  - Tugba DERE, Yozgat

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schopflocher D, Harstall C. The descriptive epidemiology of chronic pain. Chronic pain: A health policy perspective. 2008:29-40.
- [Background] Wu B, Yang L, Peng B. Ingrowth of Nociceptive Receptors into Diseased Cervical Intervertebral Disc Is Associated with Discogenic Neck Pain. Pain Med. 2019 Jun 1;20(6):1072-1077. doi: 10.1093/pm/pnz013. PMID 30848823
- [Background] Ma M, Zhang H, Liu R, Liu H, Yang X, Yin X, Chen S, Wu X. Static and Dynamic Changes of Amplitude of Low-Frequency Fluctuations in Cervical Discogenic Pain. Front Neurosci. 2020 Jul 14;14:733. doi: 10.3389/fnins.2020.00733. eCollection 2020. PMID 32760245
- [Background] Qian M, Zhao D, Qin T, Md ML, Xu H, Xu B. Increased Expression of Inflammatory Cytokines in Diseased Cervical Intervertebral Disc is Associated with Discogenic Neck Pain. 2023.
- [Background] Abdel-Aziem AA, Mohamed RR, Draz AH, Azab AR, Hegazy FA, Diab RH. The effect of McKenzie protocol vs. deep neck flexor and scapulothoracic exercises in subjects with chronic neck pain - a randomized controlled study. Eur Rev Med Pharmacol Sci. 2022 May;26(9):3138-3150. doi: 10.26355/eurrev_202205_28731. PMID 35587064
- [Background] Cuenca-Martinez F, Suso-Marti L, Sanchez-Martin D, Soria-Soria C, Serrano-Santos J, Paris-Alemany A, La Touche R, Leon-Hernandez JV. Effects of Motor Imagery and Action Observation on Lumbo-pelvic Motor Control, Trunk Muscles Strength and Level of Perceived Fatigue: A Randomized Controlled Trial. Res Q Exerc Sport. 2020 Mar;91(1):34-46. doi: 10.1080/02701367.2019.1645941. Epub 2019 Oct 18. PMID 31626568
- [Background] Southerst D, Nordin MC, Cote P, Shearer HM, Varatharajan S, Yu H, Wong JJ, Sutton DA, Randhawa KA, van der Velde GM, Mior SA, Carroll LJ, Jacobs CL, Taylor-Vaisey AL. Is exercise effective for the management of neck pain and associated disorders or whiplash-associated disorders? A systematic review by the Ontario Protocol for Traffic Injury Management (OPTIMa) Collaboration. Spine J. 2016 Dec;16(12):1503-1523. doi: 10.1016/j.spinee.2014.02.014. Epub 2014 Feb 15. PMID 24534390
- [Background] Blomgren J, Strandell E, Jull G, Vikman I, Roijezon U. Effects of deep cervical flexor training on impaired physiological functions associated with chronic neck pain: a systematic review. BMC Musculoskelet Disord. 2018 Nov 28;19(1):415. doi: 10.1186/s12891-018-2324-z. PMID 30486819
- [Background] Kang DY. Deep cervical flexor training with a pressure biofeedback unit is an effective method for maintaining neck mobility and muscular endurance in college students with forward head posture. J Phys Ther Sci. 2015 Oct;27(10):3207-10. doi: 10.1589/jpts.27.3207. Epub 2015 Oct 30. PMID 26644676
- [Background] Ganu S, Gor U. Effects of Abdominal Control Feedback and Scapular Stabilization Exercise on Chronic Neck Pain. International Journal of Health Sciences and Research. 2021;11:318-25.
- [Background] Bowering KJ, O'Connell NE, Tabor A, Catley MJ, Leake HB, Moseley GL, Stanton TR. The effects of graded motor imagery and its components on chronic pain: a systematic review and meta-analysis. J Pain. 2013 Jan;14(1):3-13. doi: 10.1016/j.jpain.2012.09.007. Epub 2012 Nov 15. PMID 23158879
- [Background] Haff GG, Triplett NT. Essentials of strength training and conditioning 4th edition: Human kinetics; 2015.
- [Background] Alghadir AH, Iqbal ZA. Effect of Deep Cervical Flexor Muscle Training Using Pressure Biofeedback on Pain and Forward Head Posture in School Teachers with Neck Pain: An Observational Study. Biomed Res Int. 2021 May 22;2021:5588580. doi: 10.1155/2021/5588580. eCollection 2021. PMID 34095302
- [Background] Neblett R, Mayer TG, Hartzell MM, Williams MJ, Gatchel RJ. The Fear-avoidance Components Scale (FACS): Development and Psychometric Evaluation of a New Measure of Pain-related Fear Avoidance. Pain Pract. 2016 Apr;16(4):435-50. doi: 10.1111/papr.12333. Epub 2015 Jul 31. PMID 26228238
- [Background] Acet N, Güzel N, Günendi Z. Nonspesifik Boyun Ağrılı Hastalarda Servikal Bölgeye Yapılan Mobilizasyonun Boyun Mobilitesiİ, Ağrı, Basınç Ağrı Eşiği ve Dizabilite Üzerine Etkisi. Gazi Sağlık Bilimleri Dergisi. 2020;5(2).
- [Background] Wand BM, Catley MJ, Rabey MI, O'Sullivan PB, O'Connell NE, Smith AJ. Disrupted Self-Perception in People With Chronic Low Back Pain. Further Evaluation of the Fremantle Back Awareness Questionnaire. J Pain. 2016 Sep;17(9):1001-12. doi: 10.1016/j.jpain.2016.06.003. Epub 2016 Jun 18. PMID 27327235
- [Background] Williams SE, Cumming J, Ntoumanis N, Nordin-Bates SM, Ramsey R, Hall C. Further validation and development of the movement imagery questionnaire. J Sport Exerc Psychol. 2012 Oct;34(5):621-46. doi: 10.1123/jsep.34.5.621. PMID 23027231
- [Background] Aytar A, Yuruk ZO, Tuzun EH, Baltaci G, Karatas M, Eker L. The Upper Extremity Functional Index (UEFI): cross-cultural adaptation, reliability, and validity of the Turkish version. J Back Musculoskelet Rehabil. 2015;28(3):489-95. doi: 10.3233/BMR-140545. PMID 25322741
- [Background] Edmondston SJ, Wallumrod ME, Macleid F, Kvamme LS, Joebges S, Brabham GC. Reliability of isometric muscle endurance tests in subjects with postural neck pain. J Manipulative Physiol Ther. 2008 Jun;31(5):348-54. doi: 10.1016/j.jmpt.2008.04.010. PMID 18558277
- [Background] Chung S, Jeong YG. Effects of the craniocervical flexion and isometric neck exercise compared in patients with chronic neck pain: A randomized controlled trial. Physiother Theory Pract. 2018 Dec;34(12):916-925. doi: 10.1080/09593985.2018.1430876. Epub 2018 Jan 24. PMID 29364754
- [Background] Domenech MA, Sizer PS, Dedrick GS, McGalliard MK, Brismee JM. The deep neck flexor endurance test: normative data scores in healthy adults. PM R. 2011 Feb;3(2):105-10. doi: 10.1016/j.pmrj.2010.10.023. PMID 21333948
- [Background] Aslan E, Karaduman A, Yakut Y, Aras B, Simsek IE, Yagly N. The cultural adaptation, reliability and validity of neck disability index in patients with neck pain: a Turkish version study. Spine (Phila Pa 1976). 2008 May 15;33(11):E362-5. doi: 10.1097/BRS.0b013e31817144e1. PMID 18469684
- [Background] Waddell G, Newton M, Henderson I, Somerville D, Main CJ. A Fear-Avoidance Beliefs Questionnaire (FABQ) and the role of fear-avoidance beliefs in chronic low back pain and disability. Pain. 1993 Feb;52(2):157-168. doi: 10.1016/0304-3959(93)90127-B. PMID 8455963
- [Derived] Dere T, Yurdakul G, Alemdaroglu-Gurbuz I. Effectiveness of motor imagery training in women with chronic neck pain: a single-blind, randomized controlled trial. Physiother Theory Pract. 2025 Dec 11:1-21. doi: 10.1080/09593985.2025.2599423. Online ahead of print. PMID 41382357